CLINICAL TRIAL: NCT00690534
Title: Insulin and Sarcopenia in the Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 05-090; 5R01AG018311 (NIH)
Record Dates: First submitted 2008-05-27; First posted 2008-06-04 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2015-01

CONDITIONS: Sarcopenia
Keywords: sarcopenia; aging; muscle metabolism
MeSH Terms: conditions — Sarcopenia | interventions — Insulin; omega-N-Methylarginine; Nitroprusside

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- CMAY (Active Comparator): Insulin in young
  Interventions: Drug: Insulin Regular
- IMAY (Experimental): L-NMMA + insulin in young
  Interventions: Drug: Insulin Regular; Drug: L-NMMA
- SNPY (Experimental): SNP in young
  Interventions: Drug: Sodium Nitroprusside
- CSNP (Active Comparator): Insulin in elderly
  Interventions: Drug: Insulin Regular
- ISNP (Experimental): SNP in elderly
  Interventions: Drug: Insulin Regular; Drug: Sodium Nitroprusside
- SNPE (Experimental): SNP in elderly
  Interventions: Drug: Sodium Nitroprusside
- CMealO (Active Comparator): Meal in elderly
  Interventions: Other: mixed meal
- SMealO (Experimental): SNP+meal in elderly
  Interventions: Drug: Sodium Nitroprusside; Other: mixed meal
- MealY (Active Comparator): meal in young
  Interventions: Other: mixed meal
- ExIns (Experimental): insulin+exercise in elderly
  Interventions: Drug: Insulin Regular
- ExMeal (Experimental): meal+exercise in elderly
  Interventions: Other: mixed meal

INTERVENTIONS:
Drug: Insulin Regular — insulin, 0.2 mU/kg/min for 3 hours
  Arms: CMAY; CSNP; ExIns; IMAY; ISNP
Drug: L-NMMA — variable rate for 3 hours
  Arms: IMAY
Drug: Sodium Nitroprusside — variable rate for 3 hours
  Arms: ISNP; SMealO; SNPE; SNPY
Other: mixed meal — mixed meal
  Arms: CMealO; ExMeal; MealY; SMealO

SUMMARY:
Muscle loss with aging is a significant contributor to disability in older people. Our general hypothesis is that loss of muscle with aging, known as sarcopenia, may be due to inability of muscle to grow in response to insulin. Our goal is to determine the mechanisms underlying this age-related insulin resistance of muscle proteins, which will allow us to define in the future specific interventions to target this defect and provide the scientific basis for the prevention and treatment of sarcopenia.

DETAILED DESCRIPTION:
Our general hypothesis is that a reduced response of muscle protein anabolism to insulin plays an important role in the loss of muscle mass with aging. Our goal is to determine the mechanisms underlying the age-related insulin resistance of muscle proteins, which will allow us to define specific interventions to target this defect and provide the scientific basis for the prevention and treatment of sarcopenia.

Our previous studies indicate that the response of muscle proteins to the anabolic action of insulin is impaired in healthy older adults as compared to younger controls, which hampers the anabolic effect of mixed feeding on muscle proteins. These changes are associated with an age-related reduction in the vasodilatory response to insulin, which, from our data, appears to be a potentially important mediator of the physiological anabolic effect of insulin on muscle proteins. Preliminary data from our laboratory also suggest that in older subjects a single bout of aerobic exercise may restore the normal response of blood flow, muscle protein synthesis and anabolism to insulin.

Therefore, we will test in healthy subjects the following specific hypotheses:

1. Insulin-induced increases in blood flow and muscle perfusion are necessary for the physiological stimulation of muscle protein synthesis and anabolism by insulin.
2. Aging reduces the vascular sensitivity to insulin, which prevents the physiological increase in blood flow and muscle perfusion in response to insulin, thereby decreasing the response of muscle protein synthesis and net balance to the anabolic action of insulin and mixed feeding.
3. Aerobic exercise can restore, in older subjects, the insulin-induced increase in blood flow and muscle perfusion to youthful levels, thus normalizing the anabolic effect of insulin and mixed feeding on muscle protein synthesis and net muscle protein balance.

We will use state-of the art stable isotope tracer techniques to measure muscle protein turnover, and a newly developed method to measure muscle perfusion in young and older subjects. The results of these studies will allow us to better define the physiological mechanisms of action of insulin on muscle protein anabolism, advance our knowledge on the pathophysiology of sarcopenia, and provide the scientific basis for the behavioral and/or pharmacological treatment of muscle loss with aging.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-40 yrs, and 65-85 yrs.
2. Ability to sign consent form (score >23 on the 30-item Mini Mental State Examination, MMSE)
3. Stable body weight for at least 3 months

Exclusion Criteria:

1. Physical dependence or frailty (impairment in any of the Activities of Daily Living (ADL), history of falls (>2/year) or significant weight loss in the past year)
2. Exercise training (>2 weekly sessions of moderate to high intensity aerobic or resistance exercise)
3. Pregnancy or nursing women.
4. Significant heart, liver, kidney, blood or respiratory disease
5. Peripheral vascular disease
6. Diabetes mellitus or other untreated endocrine disease
7. Active cancer
8. Recent (within 6 months) treatment with anabolic steroids, or corticosteroids.
9. Alcohol or drug abuse
10. Severe depression (>5 on the 15-item Geriatric Depression Scale, GDS)
11. Potential subjects who have recently donated blood in the past 60 days will be excluded from participating in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
muscle protein synthesis | 5 and 8 hours

SECONDARY OUTCOMES:
blood flow | 5 and 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Elena Volpi, MD, PhD, Principal Investigator — The University of Texas Medical Branch at Galveston
Locations (1):
- Sealy Center on Aging, University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No sharing. Drug was used off label for collection of measures for research project.

REFERENCES:
- [Result] Rasmussen BB, Fujita S, Wolfe RR, Mittendorfer B, Roy M, Rowe VL, Volpi E. Insulin resistance of muscle protein metabolism in aging. FASEB J. 2006 Apr;20(6):768-9. doi: 10.1096/fj.05-4607fje. Epub 2006 Feb 7. PMID 16464955
- [Result] Bell JA, Volpi E, Fujita S, Cadenas JG, Sheffield-Moore M, Rasmussen BB. Skeletal muscle protein anabolic response to increased energy and insulin is preserved in poorly controlled type 2 diabetes. J Nutr. 2006 May;136(5):1249-55. doi: 10.1093/jn/136.5.1249. PMID 16614412
- [Result] Bell JA, Volpi E, Fujita S, Cadenas JG, Rasmussen BB. Dysregulation of muscle fatty acid metabolism in type 2 diabetes is independent of malonyl-CoA. Diabetologia. 2006 Sep;49(9):2144-52. doi: 10.1007/s00125-006-0362-9. Epub 2006 Jul 26. PMID 16868746
- [Result] Timmerman KL, Volpi E. Amino acid metabolism and regulatory effects in aging. Curr Opin Clin Nutr Metab Care. 2008 Jan;11(1):45-9. doi: 10.1097/MCO.0b013e3282f2a592. PMID 18090658
- [Result] Fujita S, Volpi E. Amino acids and muscle loss with aging. J Nutr. 2006 Jan;136(1 Suppl):277S-80S. doi: 10.1093/jn/136.1.277S. PMID 16365098
- [Result] Dreyer HC, Volpi E. Role of protein and amino acids in the pathophysiology and treatment of sarcopenia. J Am Coll Nutr. 2005 Apr;24(2):140S-145S. doi: 10.1080/07315724.2005.10719455. PMID 15798081
- [Result] Drummond MJ, Bell JA, Fujita S, Dreyer HC, Glynn EL, Volpi E, Rasmussen BB. Amino acids are necessary for the insulin-induced activation of mTOR/S6K1 signaling and protein synthesis in healthy and insulin resistant human skeletal muscle. Clin Nutr. 2008 Jun;27(3):447-56. doi: 10.1016/j.clnu.2008.01.012. Epub 2008 Mar 14. PMID 18342407
- [Result] Drummond MJ, Dreyer HC, Pennings B, Fry CS, Dhanani S, Dillon EL, Sheffield-Moore M, Volpi E, Rasmussen BB. Skeletal muscle protein anabolic response to resistance exercise and essential amino acids is delayed with aging. J Appl Physiol (1985). 2008 May;104(5):1452-61. doi: 10.1152/japplphysiol.00021.2008. Epub 2008 Mar 6. PMID 18323467
- [Result] Fujita S, Rasmussen BB, Cadenas JG, Drummond MJ, Glynn EL, Sattler FR, Volpi E. Aerobic exercise overcomes the age-related insulin resistance of muscle protein metabolism by improving endothelial function and Akt/mammalian target of rapamycin signaling. Diabetes. 2007 Jun;56(6):1615-22. doi: 10.2337/db06-1566. Epub 2007 Mar 9. PMID 17351147
- [Result] Fujita S, Rasmussen BB, Bell JA, Cadenas JG, Volpi E. Basal muscle intracellular amino acid kinetics in women and men. Am J Physiol Endocrinol Metab. 2007 Jan;292(1):E77-83. doi: 10.1152/ajpendo.00173.2006. Epub 2006 Aug 8. PMID 16896165
- [Result] Fujita S, Rasmussen BB, Cadenas JG, Grady JJ, Volpi E. Effect of insulin on human skeletal muscle protein synthesis is modulated by insulin-induced changes in muscle blood flow and amino acid availability. Am J Physiol Endocrinol Metab. 2006 Oct;291(4):E745-54. doi: 10.1152/ajpendo.00271.2005. Epub 2006 May 16. PMID 16705054
- [Result] Bell JA, Fujita S, Volpi E, Cadenas JG, Rasmussen BB. Short-term insulin and nutritional energy provision do not stimulate muscle protein synthesis if blood amino acid availability decreases. Am J Physiol Endocrinol Metab. 2005 Dec;289(6):E999-1006. doi: 10.1152/ajpendo.00170.2005. Epub 2005 Jul 19. PMID 16030064
- [Result] Volpi E, Chinkes DL, Rasmussen BB. Sequential muscle biopsies during a 6-h tracer infusion do not affect human mixed muscle protein synthesis and muscle phenylalanine kinetics. Am J Physiol Endocrinol Metab. 2008 Oct;295(4):E959-63. doi: 10.1152/ajpendo.00671.2007. Epub 2008 Aug 19. PMID 18713956
- [Result] Drummond MJ, Miyazaki M, Dreyer HC, Pennings B, Dhanani S, Volpi E, Esser KA, Rasmussen BB. Expression of growth-related genes in young and older human skeletal muscle following an acute stimulation of protein synthesis. J Appl Physiol (1985). 2009 Apr;106(4):1403-11. doi: 10.1152/japplphysiol.90842.2008. Epub 2008 Sep 11. PMID 18787087
- [Result] Fujita S, Glynn EL, Timmerman KL, Rasmussen BB, Volpi E. Supraphysiological hyperinsulinaemia is necessary to stimulate skeletal muscle protein anabolism in older adults: evidence of a true age-related insulin resistance of muscle protein metabolism. Diabetologia. 2009 Sep;52(9):1889-98. doi: 10.1007/s00125-009-1430-8. Epub 2009 Jul 9. PMID 19588121
- [Result] Timmerman KL, Lee JL, Dreyer HC, Dhanani S, Glynn EL, Fry CS, Drummond MJ, Sheffield-Moore M, Rasmussen BB, Volpi E. Insulin stimulates human skeletal muscle protein synthesis via an indirect mechanism involving endothelial-dependent vasodilation and mammalian target of rapamycin complex 1 signaling. J Clin Endocrinol Metab. 2010 Aug;95(8):3848-57. doi: 10.1210/jc.2009-2696. Epub 2010 May 19. PMID 20484484
- [Result] Timmerman KL, Lee JL, Fujita S, Dhanani S, Dreyer HC, Fry CS, Drummond MJ, Sheffield-Moore M, Rasmussen BB, Volpi E. Pharmacological vasodilation improves insulin-stimulated muscle protein anabolism but not glucose utilization in older adults. Diabetes. 2010 Nov;59(11):2764-71. doi: 10.2337/db10-0415. Epub 2010 Aug 19. PMID 20724580
- [Result] Drummond MJ, McCarthy JJ, Sinha M, Spratt HM, Volpi E, Esser KA, Rasmussen BB. Aging and microRNA expression in human skeletal muscle: a microarray and bioinformatics analysis. Physiol Genomics. 2011 May 1;43(10):595-603. doi: 10.1152/physiolgenomics.00148.2010. Epub 2010 Sep 28. PMID 20876843
- [Result] Timmerman KL, Dhanani S, Glynn EL, Fry CS, Drummond MJ, Jennings K, Rasmussen BB, Volpi E. A moderate acute increase in physical activity enhances nutritive flow and the muscle protein anabolic response to mixed nutrient intake in older adults. Am J Clin Nutr. 2012 Jun;95(6):1403-12. doi: 10.3945/ajcn.111.020800. Epub 2012 May 9. PMID 22572647
- [Result] Drummond MJ, Dickinson JM, Fry CS, Walker DK, Gundermann DM, Reidy PT, Timmerman KL, Markofski MM, Paddon-Jones D, Rasmussen BB, Volpi E. Bed rest impairs skeletal muscle amino acid transporter expression, mTORC1 signaling, and protein synthesis in response to essential amino acids in older adults. Am J Physiol Endocrinol Metab. 2012 May 15;302(9):E1113-22. doi: 10.1152/ajpendo.00603.2011. Epub 2012 Feb 14. PMID 22338078
- [Result] Drummond MJ, Timmerman KL, Markofski MM, Walker DK, Dickinson JM, Jamaluddin M, Brasier AR, Rasmussen BB, Volpi E. Short-term bed rest increases TLR4 and IL-6 expression in skeletal muscle of older adults. Am J Physiol Regul Integr Comp Physiol. 2013 Aug 1;305(3):R216-23. doi: 10.1152/ajpregu.00072.2013. Epub 2013 Jun 12. PMID 23761639